CLINICAL TRIAL: NCT02918214
Title: Prognostic Assessment of Diastolic and Systolic Left Ventricular Function in Septic Shock
Acronym: PRODIASYS2
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Collaborators: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: I16018 (PRODIASYS2)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Septic Shock; Echocardiography; Diastolic Dysfunction; Hyperkinesia
Keywords: Septic Shock; echocardiography; diastolic dysfunction; Transthoracic; Transesophageal; hyperkinesia; prognosis
MeSH Terms: conditions — Shock, Septic; Hyperkinesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- echocardiography: Each patient will be hemodynamically assessed using echocardiography: Day1 defines the first echocardiography performed within the first 12 hours (ideally within the first 6 h) following the diagnosis of septic shock, Day2 and Day3 define the examination performed 24 to 36 h and 48 to 72 h later (guidance of treatment during the acute phase), Day end defines the examination performed after vasopressors cessation (end of hemodynamic failure). In addition, echocardiography will be performed on ICU discharge and on Day28 or on hospital discharge (whatever occurs first) to document potential reversibility of LV diastolic dysfunction. Transthoracic echocardiography will always first be performed and transesophageal echocardiography will be limited to ventilated patients without adequate surface echocardiographic image quality, under sedation and during the initial phase of septic shock (D1 to D3), according to the standards of care of participating centers.

SUMMARY:
Sepsis induces a reversible systolic and diastolic cardiac dysfunction. The presence of a left ventricular (LV) diastolic dysfunction during septic shock could favor harmful volume overload. Recently, a meta-analysis suggested a negative prognostic role of LV diastolic dysfunction in septic patients (Od Ratio: 1.82; 95%CI: 1.12 - 2.97; p = 0.02) but its external validity is hampered by the numerous limits and the heterogeneity of the studies. To date, a pathophysiological link between LV diastolic dysfunction associated with septic shock and the water balance (reflecting volume overload) remains to establish. In addition, small size studies reported an excess of mortality in patients with septic shock who were diagnosed with a high cardiac output. However, no large cohort has yet confirmed the negative prognostic role of a hyperkinetic hemodynamic profile at the initial phase of septic shock.

DETAILED DESCRIPTION:
Consecutive patients diagnosed with septic shock will be followed daily using echocardiography from Day1 (first echocardiography performed within 12h after the diagnosis of septic shock) to Day3, after vasopressor discontinuation (Day end), and on Day28 or at hospital discharge (if occurs before Day28). Echocardiographic data will be anonymized and stored in DICOM format in a dedicated database for independent measurements by an expert in echocardiography blinded from the clinical data of the patients including vital status. Vital and biological parameters usually monitored for the management of septic shock will be collected at the time of each echocardiographic assessment. Patients' vital status will be collected on Day28. The potential influence of LV diastolic dysfunction and LV hyperkinesia on prognosis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in ICU for septic shock:

  * Documented or highly suspected infection (clinically or microbiologically)
  * Causing an organ failure defined as an acute change in total SOFA score ≥ 2 points (baseline SOFA score can be assumed to be zero in the absence of pre-existing organ dysfunction)
  * And low blood pressure (sBP < 90 mmHg or a decrease of more than 40 mmHg compared to baseline, or mBP < 65 mmHg) despite a fluid loading of 30 mL/kg (except if clinical or radiological sign of pulmonary fluid overload) requiring vasopressor infusion to maintain mBP > 65 mmHg
  * And lactate level > 2 mmol/L
* Patient older than 18 years old affiliated to the French Social Security
* Non-opposition of the patient (or of its next-of-kin) to participate in the study

Exclusion Criteria:

* Ongoing dobutamine or epinephrine infusion
* Severe left valvular disease (severe stenosis, severe regurgitation ≥ grade 3)
* Constrictive pericarditis (invalidate the mitral tissue Doppler imaging)
* Pregnant women
* Patient with estimated life expectancy < 24h.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in the ICU but also in Emergency Departments if they present with septic shock before ICU admission
Sampling Method: Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Survival | Day 28
  Survival at one month

SECONDARY OUTCOMES:
Daily water balance | Day 1 to Day 3
  The daily water balance (from Day1 to Day3 included) will be measured
Cumulated water balances | Day 4
  The cumulated water balance on Day4 (sum of water balances recorded from Day1 to Day3 included) will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Marine GOUDELIN, MD, Principal Investigator — University Hospital, Limoges
Locations (10):
- France (10):
  - University Hospital, Amiens
  - University Hospital, Brest
  - University Hospital, Limoges
  - CHU de Nancy, Nancy
  - CH d'Orleans, Orléans
  - Aphp - Ambroise Paré, Paris
  - CHU de Poitiers, Poitiers
  - Felix Guyon Hospital, Saint-Denis
  - University Hospital, Toulouse
  - University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vignon P, Charron C, Legras A, Musset F, Slama M, Prat G, Silva S, Vandroux D, Muller G, Levy B, Boissier F, Evrard B, Goudelin M, Mankikian S, Nay MA, Jabot J, Riu B, Bailly P, Maizel J, Leger J, Vieillard-Baron A; CRICS-TRIGGERSEP Network. Left ventricular diastolic dysfunction is prevalent but not associated with mortality in patients with septic shock. Intensive Care Med. 2025 Jan;51(1):94-105. doi: 10.1007/s00134-024-07748-2. Epub 2025 Jan 7. PMID 39774865